CLINICAL TRIAL: NCT02841787
Title: Technology Assisted Intervention for the Treatment and Prevention of Depression
Brief Title: Online Peer Networked Collaborative Learning for Managing Depressive Symptoms
Acronym: MoodTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P20MH090318-FT; P20MH090318 (NIH); NCT01912664 (obsolete NCT alias)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: Depression; Web-based intervention; Aging; Geriatrics; Social network; Older adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individual Internet Intervention (III) (Experimental): Coached internet intervention based on the principles of cognitive behavioral therapy (CBT) for depressed older adults delivered individually by 2 clinical psychologists.
  (iCBT for late life depression without social network included.)
  Interventions: Behavioral: iCBT for late life depression
- Internet Intervention+Peer Supp.(II+PS) (Experimental): Coached internet intervention based on the principles of cognitive behavioral therapy (CBT) for depressed older adults delivered with peer support; group moderation was provided by 2 clinical psychologists.
  (iCBT for late life depression with social network included.)
  Interventions: Behavioral: iCBT for late life depression
- Waitlist Control (WLC) (No Intervention): Waiting period, no intervention administered. WLC participants received access to the III following the 8-week waiting period.

INTERVENTIONS:
Behavioral: iCBT for late life depression
  Arms: Individual Internet Intervention (III); Internet Intervention+Peer Supp.(II+PS)

SUMMARY:
The goal of this field trial is to tailor and test a web-based intervention in adults 65 years of age or older. Two versions of the web-based intervention have been created and will be tested--one with an online social network and one without an online social network. The purpose of this study is to: pilot a novel intervention, examine methods to improve adherence to web-based interventions (e.g., peer network); collect data on feasibility, acceptability, and efficacy of an web-based intervention for late life depression; and ultimately, to overcome the numerous barriers to treating depression in later life.

ELIGIBILITY:
Inclusion Criteria:

* Has elevated depressive symptoms
* Has a telephone, e-mail account, computer, and broadband access to the Internet.
* Has basic internet skills and is able to access the internet independently
* Is able to speak and read English.
* Is at least 65 years of age.
* Is able to give informed consent.

Exclusion Criteria:

* Has hearing or voice impairment that would prevent participation in psychotherapy
* Has visual impairment that would prevent completion of assessment materials.
* Is diagnosed with a psychotic disorder, bipolar disorder, dissociative disorder, current substance abuse, or other diagnosis for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous.
* Is currently receiving individual psychotherapy or planning to receive psychotherapy during the 8-week treatment phase of the study
* Is planning to be out of town or unavailable for an extended period of time during the study without access to the Internet
* Exhibits severe suicidality, including ideation, plan, and intent.
* Has initiated treatment with an antidepressant in past 14 days. Once patients have been on a stable dose for 14 days and do not have an appointment with a physician or psychiatrist to change this dose, the patient will be eligible based on this criterion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Individual Internet Intervention (III): Coached internet intervention based on the principles of cognitive behavioral therapy (CBT) for depressed older adults delivered individually by 2 clinical psychologists.
- Internet Intervention With Peer Support (II+PS): Coached internet intervention based on the principles of cognitive behavioral therapy (CBT) for depressed older adults delivered with peer support; group moderation was provided by 2 clinical psychologists.
- Waitlist Control (WLC): WLC participants received access to the III following the 8-week waiting period.
Period: Overall Study
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS) | Waitlist Control (WLC)
Started | 12 | 23 | 12
Completed | 9 | 19 | 12
Not Completed | 3 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Symptoms dropped below threshold | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS) | Waitlist Control (WLC) | Total
Number analyzed (Participants) | 12 | 23 | 12 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (3.4) | 69.5 (4.3) | 70 (4.7) | 69.6 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 8 | 32
  Male | 4 | 7 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 22 | 12 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 11 | 19 | 11 | 41
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 1
Annual gross household income (x1000) [Median (Inter-Quartile Range); unit: USD] | 37.5 [33 to 45] | 37 [22.2 to 50] | 50 [34 to 115] | 41 [29 to 50]
Marital Status [Count of Participants; unit: Participants]
  No Partner | 8 | 16 | 5 | 29
  Partner | 4 | 7 | 7 | 18
Education [Count of Participants; unit: Participants]
  Some High School | 0 | 0 | 1 | 1
  Some College | 1 | 5 | 1 | 7
  2-yr College (Associate's) | 0 | 5 | 2 | 7
  4-yr College (Bachelor's) | 3 | 6 | 4 | 13
  Master's Degree | 5 | 5 | 2 | 12
  Doctoral Degree (PhD, MD, JD) | 3 | 2 | 2 | 7
Employment Status [Count of Participants; unit: Participants]
  Employed | 3 | 4 | 3 | 10
  Retired | 9 | 18 | 7 | 34
  Unemployed/Disability | 0 | 1 | 2 | 3
Health Insurance [Count of Participants; unit: Participants]
  Insured | 12 | 22 | 12 | 46
  Medicare | 10 | 19 | 11 | 40
  Medicaid | 1 | 3 | 0 | 4
Taking antidepressant medication [Count of Participants; unit: Participants]
  No | 7 | 18 | 7 | 32
  Yes | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire - 9 (PHQ-9) - Depression Severity Module
Description: The PHQ-9 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-27. Higher values represent a worse outcome. Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-27 is severe.
  The data table below shows PHQ-9 pre- and post- intervention score differences by group.
Time Frame: Baseline and Week 8 - Difference in PHQ-9 score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS) | Waitlist Control (WLC)
Number analyzed (Participants) | 9 | 19 | 12
units on a scale | -5.4 (2.4) | -4.8 (4.4) | -1.1 (4.7)
Statistical Analysis 1: Comparison: Individual Internet Intervention (III); Test type: Superiority; p < .001, t-test, 2 sided — The threshold for significance was alpha=0.05
Statistical Analysis 2: Comparison: Internet Intervention With Peer Support (II+PS); Test type: Superiority; p < .001, t-test, 2 sided — The threshold for significance was alpha=0.05
Statistical Analysis 3: Comparison: Waitlist Control (WLC); Test type: Superiority; p = 0.44, t-test, 2 sided — The threshold for significance was alpha=0.05
Statistical Analysis 4: Comparison: Individual Internet Intervention (III) vs Internet Intervention With Peer Support (II+PS) vs Waitlist Control (WLC); Test type: Superiority; p = 0.03, ANOVA — The threshold for significance was alpha=0.05
Statistical Analysis 5: Comparison: Individual Internet Intervention (III) vs Internet Intervention With Peer Support (II+PS); Test type: Superiority; p = 0.68, t-test, 2 sided — The threshold for significance was alpha=0.05
Statistical Analysis 6: Comparison: Individual Internet Intervention (III) vs Waitlist Control (WLC); Test type: Superiority; p = 0.02, t-test, 2 sided — The threshold for significance was alpha=0.05
Statistical Analysis 7: Comparison: Internet Intervention With Peer Support (II+PS) vs Waitlist Control (WLC); Test type: Superiority; p = 0.03, t-test, 2 sided — The threshold for significance was alpha=0.05

2. Primary Outcome: Mean Number of Sessions Across the 8-week Trial
Time Frame: 8 weeks
Population: Out of the 12 participants who started Individual Internet Intervention, one participant was administratively dropped (no longer eligible for the study) before treatment started; only 11 participants were analyzed.
Measure: Mean (Standard Deviation); unit: number of sessions
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS)
Number analyzed (Participants) | 11 | 23
number of sessions | 45.6 (24.9) | 49.1 (35.8)

3. Primary Outcome: System Usability Scale (SUS)
Description: The System Usability Scale (SUS) is a usability scale that can be used for global assessments of systems usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Originally created by John Brooke in 1986, it allows you to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. A SUS score above a 68 would be considered above average and anything below 68 is below average.
Time Frame: Week 8
Population: Participants were included in outcome analyses if they completed assessments at both baseline and week 8; for the Individual Internet Intervention (III) arm, 9 participants met this criterion, and for Internet Intervention with Peer Support (II+PS), 21 participants met this criterion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS)
Number analyzed (Participants) | 9 | 21
units on a scale | 68.75 (16.09) | 60.5 (16.69)

4. Primary Outcome: Average Coaching Time Per Participant by Group
Description: The average time spent on messages and calls and on group moderation.
Time Frame: 8 weeks
Population: Participants were included in outcome analyses if they completed assessments at both baseline and week 8; for the Individual Internet Intervention (III) arm, 9 participants met this criterion, and for Internet Intervention with Peer Support (II+PS), 19 participants met this criterion.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS)
Number analyzed (Participants) | 9 | 19
Minutes | 134.33 (28.43) | 92.43 (32.36)
Statistical Analysis 1: Comparison: Individual Internet Intervention (III) vs Internet Intervention With Peer Support (II+PS); Test type: Superiority; p = 0.003, t-test, 2 sided — The threshold for significance was alpha=0.05

ADVERSE EVENTS:
Time Frame: 8 months (January 2016 through September 2016)
Arm/Group | Individual Internet Intervention (III) | Internet Intervention With Peer Support (II+PS) | Waitlist Control (WLC)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/23 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/23 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/23 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes